CLINICAL TRIAL: NCT05633563
Title: The Effect of Trimetazidine on Mitochondrial Function, Myocardial Performance, and Invasive Hemodynamics in Patients Diagnosed With Wild-Type Transthyretin Cardiac Amyloidosis
Acronym: CACTuS - TMZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, PhD, DMSci, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 72864
Record Dates: First submitted 2021-10-15; First posted 2022-12-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Transthyretin Amyloid Cardiopathy; Mitochondrial Pathology
MeSH Terms: interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Drug (Active Comparator): Study participants receiving Trimetazidine
  Interventions: Drug: Trimetazidine
- Placebo (Placebo Comparator): Study participants receiving placebo (calcium)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimetazidine — Oral intake of capsules
  Arms: Active Drug
Drug: Placebo — Oral intake of capsules
  Arms: Placebo

SUMMARY:
Wild-type transthyretin cardiac amyloidosis (ATTRwt) is a deposition disorder in which one of the proteins of the body misfolds and accumulates at various places in the body, including the heart, leading to both mechanical and cellular damage. The gradual development of the disease will ultimately lead to heart failure and death

The protein which deposits in the heart of patients, damages both the heart mechanically as the myocardium becomes rigid and hypertrophic over time but also at the cellular level. Cell damage can be observed by elevated blood tests for cell damage (Troponin) and during exercise tests that show patients' hearts burning oxygen inefficiently when exposed to physical stress compared with the hearts of healthy individuals . No one has, however, intimately studied this cellular damage.

Vastarel® (Trimetazidine, TMZ) is an already known drug for the treatment of chest pain. The mechanism of action indicates that it may have an effect on patients with cardiac amyloidosis.

The study aims to investigate the effects of TMZ on the mitochondrial function, myocardial performance, and invasive hemodynamics in patients with ATTRwt with a randomized, double-blinded, crossover-trial.

ELIGIBILITY:
Inclusion Criteria:

* Wild-type transthyretin cardiac amyloidosis
* NAC stage I
* NYHA class of I or II
* Informed consent

Exclusion Criteria:

* Other, similar diagnoses
* Hereditary transthyretin cardiac amyloidosis
* Light chain amyloidosis
* Morbus Waldenstrøm
* Myelomatosis
* Medical treatment with loop diuretics in standard doses (40 mgx1 daily)
* Contraindications to trimetazidine
* Significant comorbidity assessed by the investigators
* Unable to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change: pulmonary capillary wedge pressure (PCWP) | Four weeks of treatment
  We hypothesize a change in PCWP of 5 mmHg between the active drug and placebo using right heart catheterization.

SECONDARY OUTCOMES:
Change: cardiac index (CI) | Four weeks of treatment
  We hypothesize a change in CI of 0.5 L/min between the active drug and placebo using right heart catheterization.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Aarhus N, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided